CLINICAL TRIAL: NCT04079998
Title: A Prospective, Randomized, Controlled Study to Determine the Superiority of a Fabric-based Wireless Electroceutical Dressing, Procellera® Compared to Standard of Care Treatment in Mitigating Biofilm Formation in Acute Trauma and Burn Wounds
Brief Title: Procellera® Compared to Standard of Care Treatment in Mitigating Biofilm Formation in Acute Trauma and Burn Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2018.065
Record Dates: First submitted 2019-03-27; First posted 2019-09-06 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Trauma-related Wound; Burn, Partial Thickness
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will have two wound sites that will be randomized to receive either the standard of care treatment or the Procellera® (electroceutical) dressing.
Who Masked: Outcomes Assessor
Masking Description: Biopsies obtained will be sent to Indiana University for blinded processing and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Procellera® dressing (Experimental): The Procellera® dressing will be applied to the wound site after standard of care cleaning and debridement. The dressing will be maintained according to the manufacturer's instructions for use.
  Interventions: Device: Procellera®
- Standard of Care (Active Comparator): The Standard of care as prescribed will be followed for the dressing application for the wound site. Dressings will be applied to the wound site after standard of care cleaning and debridement.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Procellera® — Application of Procellera® dressing.
  Arms: Procellera® dressing
Other: Standard of Care — Application of standard of care dressings as prescribed.
  Arms: Standard of Care

SUMMARY:
The objective of the study is to evaluate Procellera® , a novel FDA approved antimicrobial wound dressing in a prospective, randomized, controlled clinical study. The hypothesis is that when the dressing is moistened, the low electric field created by moisture-activated elemental silver and zinc electro-couple will prevent formation of biofilm in wounds or to disrupt existing biofilm.

DETAILED DESCRIPTION:
The healing of traumatic wounds, to include burns, can be compromised by the presence of infection so efforts are made to prevent or diagnose infection early in order to mitigate the negative impact on healing. Electric stimulation has previously been shown to have both bacteriostatic and bactericidal effects in wounds. Until now, administering low intensity electric field/micro-current as a therapy to mitigate biofilm infection and to improve wound healing was not feasible. In this study the investigators will use Procellera® , a FDA approved fabric based wireless electroceutical dressing (WED) consisting of a silver-zinc electro-couple for the prevention of wound biofilm formation. The dressing generates a low electric field (~1V) upon activation by a moist environment, which mitigates biofilm formation and promotes wound healing. The objectives of the study are to evaluate the efficacy of a wireless electroceutical dressing to prevent the formation or disrupting existing biofilms. The investigators will conduct a prospective, randomized controlled clinical trial using the Procellera® dressing compared to the standard of care. Treatment sites will be randomized to either receiving Procellera® or the standard of care treatment. Objective measurements and assessments will be completed during subject follow-up visits for up to one month post treatment. This includes biopsies to calculate bacterial load by assessing colony forming unit (CFU) count and bacterial film visualization using scanning electron microscopy, histology, clinical assessment of infection, Transepidermal Water Loss (TEWL) and wound photography.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Willing and able to provide informed consent
* Participant has acute partial-thickness or full-thickness wounds caused by trauma or partial-thickness burns that are ≥ 300 cm2 in size in one contiguous area or two separate wound sites ≥ 150 cm2 each

Exclusion Criteria:

* Pregnancy
* Prisoner
* Active malignancy or immunosuppressive therapy
* Current systemic steroid use
* Known allergy or sensitivity to silver or zinc
* Participant's proposed study wound site has any of the following conditions:
* Location is on the hands, face or feet
* Full-thickness burn wounds
* Exposure of visceral organs
* Exposure of hardware or prosthetic exposure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Presence of biofilm | Day seven
  Presence of biofilm will be assessed by obtaining a wound biopsy and analyzing with Scanning Electron Microscopy.
Rate of eradication of biofilm production | Day 7
  Presence of biofilm will be assessed by obtaining a wound biopsy and analyzing with Scanning Electron Microscopy.

SECONDARY OUTCOMES:
Incidence of infection | Day 0-30
  Wounds will be assessed for the presence of clinical evidence indicating infection.
Percent epithelialization | Day 7
  The percentage of epitheliazation will be assessed utilizing clinical assessments and the Silhouette Star wound camera.
Quality of healing | Day 30
  Quality of healing post-epithelialization as measured by the validated Patient Observer Scar Assessment Scale (POSAS)
Quantitative bacterial load calculation | Day 7
  Quantitative bacterial load will be assessed by obtaining a wound biopsy and analyzed by performing colony forming unit counts
Incidence of adverse events | Day 0-30
  The incidence of adverse events will be reported to assess safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan RK, Nuutila K, Mathew-Steiner SS, Diaz V, Anselmo K, Batchinsky M, Carlsson A, Ghosh N, Sen CK, Roy S. A Prospective, Randomized, Controlled Study to Evaluate the Effectiveness of a Fabric-Based Wireless Electroceutical Dressing Compared to Standard-of-Care Treatment Against Acute Trauma and Burn Wound Biofilm Infection. Adv Wound Care (New Rochelle). 2024 Jan;13(1):1-13. doi: 10.1089/wound.2023.0007. Epub 2023 Apr 11. PMID 36855334